CLINICAL TRIAL: NCT04291391
Title: The Alberta NutrIMM (Nutrition and Immune Function) Study: Establishing the Importance of Diet and Insulin Resistance in Modulating Immune Function in Obesity
Brief Title: The Alberta NutrIMM Study - Nutrition and Immunity
Acronym: NutrIMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00085839
Record Dates: First submitted 2019-11-29; First posted 2020-03-02 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
Keywords: inflammation; diabetes; obesity; lean
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Inflammation; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: 4-parallel arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Individuals without obesity and normoglycemia (NG) (Lean-NG) (Experimental): Those assigned to the Lean-NG group will receive a North American-type diet diet for 4 weeks.
  Interventions: Other: North American-type diet
- Individuals with obesity and NG (Obese-NG) (Experimental): Those assigned to the Obese-NG group will receive a North American-type diet diet for 4 weeks.
  Interventions: Other: North American-type diet
- Individuals with obesity and glucose intolerance (GI) (Obese-GI) (Experimental): Those assigned to the Obese-GI group will receive a North American-type diet diet for 4 weeks.
  Interventions: Other: North American-type diet
- Individuals with obesity and type 2 diabetes (T2D) (Obese-T2D) (Experimental): Those assigned to the Obese-T2D group will receive a North American-type diet diet for 4 weeks.
  Interventions: Other: North American-type diet

INTERVENTIONS:
Other: North American-type diet — All groups will receive an isocaloric diet for 4 weeks composed of 48% of energy as carbohydrate, 17% as protein, and 35% as lipid (12.5% of saturated fat, 13% of monounsaturated fat, and 6% of polyunsaturated fat), designed to reflect as closely as possible current macronutrient intake averages in North America/Canada.America/Canada (35% of energy as fat, 12.5% as saturated fat, 13% as monounsaturated fat, 6% as polyunsaturated fat, 48% as carbohydrate, 17% as protein)

SUMMARY:
This study will investigate the effect of body weight, diet, and high blood sugar levels, under controlled feeding conditions, on immune function in individuals with and without obesity.

This study will be a non-randomized, four-arm parallel group, clinical trial under controlled feeding conditions (4-week nutritional intervention using a North American-type diet). A sample size of n=128 participants will be allocated into one of the following groups:

* Individuals without obesity and normoglycemia (NG) (Lean-NG)
* Individuals with obesity and normoglycemia (Obese-NG)
* Individuals with obesity and glucose intolerance (GI) (Obese-GI)
* Individuals with obesity and type 2 diabetes (T2D) (Obese-T2D)

The following outcomes will be analyzed:

* Immune cell function (ex-vivo cytokine production after stimulation with mitogen and T cell proliferation);
* Immune cell phenotypes;
* Systemic inflammation (C-reactive protein and plasma cytokines);
* Glucose, insulin, glycated hemoglobin (HbA1c), and lipids;
* Fatty acids and phospholipds composition in plasma and red blood cells membrane.

ELIGIBILITY:
Inclusion Criteria

* Age of 18 years to 70 years;
* Body weight stable (± 3%) for at least three months prior to study commencement;
* Body mass index (1) between 18.5 and 24.9 (± 0.5) kg/m2 or (2) between 30 and 50 kg/m2 (± 0.5) kg/m2 or waist circumference >88 cm or > 102 cm for females and males, respectively;

See below for specific group allocation criteria based on glucose, HbA1c, High density lipoprotein cholesterol (HDL-C), and triglycerides.

* Fasting blood glucose levels (mmol/L): < 5.6 (Lean-NG and Obese-NG), 5.6-6.9 (Obese-GI), and ≥ 7.0 (Obese-T2D);
* HbA1c (%): < 5.5 (Lean-NG and Obese-NG), 5.5-6.4 (Obese-GI), and ≥ 6.5 (Obese-T2D);
* Blood Pressure (mmHg): < 130/85 (Lean-NG and Obese-NG), not required for Obese-GI and Obese-T2D;
* Triglycerides (mmol/L): < 1.7 (Lean-NG and Obese-NG), not required for Obese-GI and Obese-T2D;
* HDL-C (mmol/L): ≥ 1.03 for males and ≥ 1.29 for females (Lean-NG and Obese-NG), not required for Obese-GI and Obese-T2D.

Exclusion Criteria

* Current or recent history cardiovascular diseases or events (e.g., ischemic, rheumatic, or congenital heart disease, stroke, peripheral vascular disease, heart failure, familial hypercholesterolemia or other monogenic dyslipidemia), use of cardiac implantable electronic devices;
* Current or recent cancer, including remission, during the last five years;
* Diseases known to affect the immune system, such as infectious, inflammatory, and autoimmune diseases or autoimmune-related or suspected conditions (e.g., T1D, systemic lupus erythematosus, inflammatory bowel disease), except for psoriasis, atopic dermatitis, and rheumatoid arthritis. Continuous use of anti-inflammatory or immunosuppressant drugs and supplements for which washout is not possible, except for medications which participants with obesity could not refrain from (e.g., baby aspirins);
* Renal disorders, endocrine disorders other than T2D (e.g., acromegaly, Addison's disease, Cushing's disease);
* Untreated or uncontrolled thyroid diseases (e.g., Hashimoto's disease, hypothyroidism, hyperthyroidism);
* Known allergy, aversion to any components of the menu, or restricted dietary patterns (e.g., gluten-free diet, vegetarianism, kosher or halal diets) for which accommodations within the menu are not possible;
* Participants under titration of their medication or initiating a new treatment or HbA1c >10.5%;
* Women who are pregnant or plan to become pregnant during the study duration, who are lactating, who have an irregular menstrual cycle or are in perimenopause;
* Regular use of cannabis (e.g. smoking);
* Taking part in any other intervention study that might affect the outcomes of the current study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Differences between groups in IL-2 Secretion by Peripheral Blood Mononuclear Cells (PBMC) After Ex-vivo Stimulation with Phytohemagglutinin (PHA) at Week 4 | Week 4
  PBMCs will be stimulated with PHA for 48h and IL-2 will be quantified using enzyme-linked immunosorbent assay (ELISA).
Differences between groups in circulating C-reactive protein (CRP) at Week 4 | Week 4
  CRP will be measured by Alberta Precision Labs using an immunoturbidimetric assay

SECONDARY OUTCOMES:
Change from Baseline in IL-2 Secretion by PBMC After Ex-vivo Stimulation with mitogens at Week 4 and Differences Between Groups at Baseline and Week 4 | Baseline and Week 4
  PBMCs will be stimulated with Pokeweed Mitogen (PWM) and Phorbol Myristate Acetate and Ionomycin (PMAi), for 48h and IL-2 will be quantified using ELISA
Change from Baseline in IL-1B Secretion by PBMC After Ex-vivo Stimulation with mitogens at Week 4 and Differences Between Groups at Baseline and Week 4 | Baseline and Week 4
  PBMCs will be stimulated with Lipopolysaccharides (LPS) and PWM for 48h and PBMCs will be stimulated with PHA, LPS, PWM, and PMAi for 48h and IFN-y will be quantified using ELISA
Change from Baseline in IFN-y Secretion by PBMC After Ex-vivo Stimulation with mitogens at Week 4 and Differences Between Groups at Baseline and Week 4 | Baseline and Week 4
  PBMCs will be stimulated with PHA, LPS, PWM, and PMAi for 48h and IFN-y will be quantified using ELISA
Change from Baseline in TNF-a Secretion by PBMC After Ex-vivo Stimulation with mitogens at Week 4 and Differences Between Groups at Baseline and Week 4. | Baseline and Week 4
  PBMCs will be stimulated with PHA, LPS, PWM, and PMAi for 48h and TNF-a will be quantified using ELISA
Change from Baseline in IL-10 Secretion by PBMC After Ex-vivo Stimulation with mitogens at Week 4 and Differences Between Groups at Baseline and Week 4 | Baseline and Week 4
  PBMCs will be stimulated with PHA, LPS, PWM, and PMAi for 48h and IL-10 will be quantified using ELISA
Change from Baseline in IL-6 Secretion by PBMC After Ex-vivo Stimulation with mitogens at Week 4 and Differences Between Groups at Baseline and Week 4 | Baseline and Week 4
  PBMCs will be stimulated with PHA, LPS, PWM, PMAi for 48h and IL-6 will be quantified using ELISA
Change from Baseline in T cell proliferation at Week 4 and Differences Between Groups at Baseline and Week 4 | Baseline and Week 4
  PBMCs will be stimulated with anti-CD3/anti-CD28 for 72h and proliferation will be quantified using alamarBlue dye method, which is a reliable and sensitive assay
Change from Baseline in T Cells at Week 4 and Differences Between Groups at Baseline and Week 4 | Baseline and Week 4
  Immune cell phenotype of T cells will be determined using immunofluorescence staining for flow cytometry. The following monoclonal antibodies will be used: CD3, CD4, CD8, CD25, CD28, CD45RA, CD45RO, CTLA-4 (CD152), CD192, FoxP3, CD183, CD194, CCR10, CD196, and CD185. Data visualization will be performed in FlowJo software
Change from Baseline in B Cells at Week 4 and Differences Between Groups at Baseline and Week 4 | Baseline and Week 4
  Immune cell phenotype of B cells will be determined using immunofluorescence staining for flow cytometry. The following monoclonal antibodies will be used: CD19, CD20, ICAM-1 (CD54), CD80, and CD192. Data visualization will be performed in FlowJo software.
Change from Baseline in Dendritic Cells at Week 4 and Differences Between Groups at Baseline and Week 4 | Baseline and Week 4
  Immune cell phenotype of dendritic cells will be determined using immunofluorescence staining for flow cytometry. The following monoclonal antibodies will be used: CD11c, CD80, CD213, CD273, and HLA-DR. Data visualization will be performed in FlowJo software
Change from Baseline in Natural Killer Cells at Week 4 and Differences Between Groups at Baseline and Week 4 | Baseline and Week 4
  Immune cell phenotype of T cells will be determined using immunofluorescence staining for flow cytometry. The following monoclonal antibodies will be used: CD3, CD16, and CD56. Data visualization will be performed in FlowJo software
Change from Baseline in Monocytes at Week 4 and Differences Between Groups at Baseline and Week 4 | Baseline and Week 4
  Immune cell phenotype of Monocytes will be determined using immunofluorescence staining for flow cytometry. The following monoclonal antibodies will be used: CD11c, CD14, ICAM-1 (CD54), CD80, CD86, CD273, and HLA-DR. Data visualization will be performed in FlowJo software
Change from Baseline in IL-6 Concentrations at Week 4 and Differences Between Groups at Baseline and Week 4. | Baseline and Week 4
  IL-6 will be quantified using a multiplex assay (mesoscale).
Change from Baseline in TNF-a Concentrations at Week 4 and Differences Between Groups at Baseline and Week 4. | Baseline and Week 4
  TNF-a will be quantified using a multiplex assay (mesoscale).
Change from Baseline in Complete Blood Cell Count and Differential at Week 4 and Differences Between Groups at Baseline and Week 4 | Baseline and Week 4
  Blood count and differential will be analyzed by Alberta Precision Labs in whole blood by fluorescent flow cytometry using a semi-conductor laser and hydrodynamic focusing in dedicated channels using an automated hematology analyzer
Change from Baseline in Circulating Glucose Levels at Week 4 and Differences Between Groups at Baseline and Week 4 | Baseline and Week 4
  Glucose will be measured by Alberta Precision Labs with an UV testing using an enzymatic reference method with hexokinase
Change from Baseline in Circulating Insulin Levels at Week 4 and Differences Between Groups at Baseline and Week 4 | Baseline and Week 4
  Insulin will be measured by Alberta Precision Labs using an electrochemiluminescence immunoassay
Change from Baseline in Circulating Hemoglobin A1c Levels at Week 4 and Differences Between Groups at Baseline and Week 4 | Baseline and Week 4
  HbA1c will be measured by Alberta Precision Labs using a turbidimetric inhibition immunoassay for hemolyzed whole blood
Change from Baseline in Circulating Triglycerides Levels at Week 4 and Differences Between Groups at Baseline and Week 4 | Baseline and Week 4
  Triglycerides will be measured by Alberta Precision Labs using an enzymatic colorimetric assay
Change from Baseline in Circulating Total Cholesterol Levels at Week 4 and Differences Between Groups at Baseline and Week 4 | Baseline and Week 4
  Total Cholesterol will be measured by Alberta Precision Labs using an enzymatic colorimetric assay
Change from Baseline in Circulating Low-Density Lipoprotein Cholesterol Levels at Week 4 and Differences Between Groups at Baseline and Week 4 | Baseline and Week 4
  LDL-C is calculated using the following equation: [Total cholesterol - HDLc - (Triglycerides/2.2)]
Change from Baseline in Circulating High-Density Lipoprotein Cholesterol Levels at Week 4 and Differences Between Groups at Baseline and Week 4 | Baseline and Week 4
  High-Density Lipoprotein Cholesterol will be measured by Alberta Precision Labs using an enzymatic colorimetric assay
Change from Baseline in Circulating Non-High Density Lipoprotein Cholesterol Levels at Week 4 and Differences Between Groups at Baseline and Week 4 | Baseline and Week 4
  Non-HDL c is derived from the calculation of total cholesterol minus HDL-c
Differences Between Groups at Week 4 in Circulating Glucose Levels before and after an Oral Glucose Tolerance Test | Week 4
  Blood will be collected at the following time points after consuming the glucose solution: 0, 30, 60, 90, 120, 150, and 180 minutes. Plasma glucose concentrations will be measured using the hexokinase/glucose-6-phosphate dehydrogenase method using a clinical chemistry analyzer
Change from Baseline in Total Lipids Fatty Acids Composition in Plasma and Red Blood Cells at Week 4 and Differences Between Groups at Baseline and Week 4 | Baseline and Week 4
  Proportion of fatty acids will be determined using gas chromatography
Change from Baseline in Phospholipids Fatty Acids Composition in Red Blood Cells at Week 4 and Differences Between Groups at Baseline and Week 4. | Baseline and Week 4
  Proportion of fatty acids from phospholipids will be determined using gas chromatography
Change from Baseline in Phospholipids Classes Quantifications in Red Blood Cells at Week 4 and Differences Between Groups at Baseline and Week 4. | Baseline and Week 4
  Quantification of phospholipds will be determined by high performance liquid chromatography

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Richard, PhD, RD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Braga Tibaes JR, Barreto Silva MI, Azarcoya-Barrera J, Blanco Cervantes P, Makarowski A, Mereu L, Richard C. Assessment of immune function in individuals without and with obesity and normoglycemia, glucose intolerance, or type 2 diabetes: primary findings of the NutrIMM study, a single-arm controlled feeding trial. Am J Clin Nutr. 2025 Jun;121(6):1315-1327. doi: 10.1016/j.ajcnut.2025.03.003. Epub 2025 Apr 22. PMID 40467164
- [Derived] Braga Tibaes JR, Barreto Silva MI, Makarowski A, Cervantes PB, Richard C. The nutrition and immunity (nutrIMM) study: protocol for a non-randomized, four-arm parallel-group, controlled feeding trial investigating immune function in obesity and type 2 diabetes. Front Nutr. 2023 Sep 1;10:1243359. doi: 10.3389/fnut.2023.1243359. eCollection 2023. PMID 37727636